CLINICAL TRIAL: NCT00617396
Title: An Open Label Study of Seroquel SR® (Quetiapine) for the Treatment of Refractory and Treatment Resistant Functional Bowel Disorders
Brief Title: Open Label Seroquel (Quetiapine) Study for Treatment Resistant Functional Bowel Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRUSQUET0448
Record Dates: First submitted 2008-02-05; First posted 2008-02-18 (Estimated); Results first posted 2014-03-21 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2014-02

CONDITIONS: Functional Bowel Disorders
Keywords: Irritable Bowel Syndrome; Seroquel; Abdominal Pain
MeSH Terms: conditions — Irritable Bowel Syndrome; Abdominal Pain | interventions — Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Quetiapine treatment group (Experimental): All subjects will receive seroquel treatment for 8 weeks. Seroquel is the intervention.
  Interventions: Drug: Quetiapine (50 mg/day-100mg/day)

INTERVENTIONS:
Drug: Quetiapine (50 mg/day-100mg/day) — Subject begin with a dose quetiapine of 50mg for 2 weeks, increasing to 100mgs for the remainder of the study. (8 weeks total)
  Other Names: Seroquel

SUMMARY:
Purpose: We are proposing to examine, via open label trial, the use of Seroquel® for patients with moderate to severe functional bowel symptoms who are not receiving adequate relief from their symptoms on their present regimen of SNRI or TCA antidepressant agents.

Participants: Primary eligibility will be determined of patients at The UNC Center for Functional GI & Motility Disorders Clinic who score in the moderate to severe range on the Functional Bowel Disorders Severity Index (FBDSI ≥ 37) who have failed or have incomplete treatment responses of medications including at least one prior trial of antidepressant medication.

Procedures (methods): We will monitor several patient and symptom related outcomes, as well as evaluate health related quality of life, psychological distress and related psychosocial measures to determine if the addition of Seroquel® over and above the use of an antidepressant improves clinical response based on an adequate relief measure as well as selected secondary outcomes. We will also determine when treatment benefit is related to effects on pain, the associated psychological co-morbidities seen in this population, or both factors.

DETAILED DESCRIPTION:
The UNC Center for Functional GI & Motility Disorders Clinic frequently receives referrals for patients with chronic and treatment refractory symptoms of abdominal pain and bowel dysfunction. Many of these patients are diagnosed with irritable bowel syndrome, painful functional constipation or functional abdominal pain syndrome using Rome III criteria. The presenting symptoms of the referral population are frequently in the severe range, with patients having intensely painful symptoms, Axis I and Axis II co-morbidities, and impaired health related quality of life. Failure of multiple standard treatment attempts prior to referral is customary for patients seen in our clinic. Additionally, a greater number of patients only experience a partial response to standard treatment. We are therefore attempting to address these patients utilizing novel treatment strategies such as we propose here.

ELIGIBILITY:
Inclusion Criteria:

* The subject has been diagnosed with a painful functional bowel disorder lasting longer than six months
* The subject achieves a score greater than 37 on the Functional Bowel Disorders Severity Index
* Four weeks on anti-depressant medications did not lead to adequate relief of the GI symptoms

Exclusion Criteria:

* Patients who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others
* Known intolerance or lack of response to Seroquel as judged by the investigator
* Use of prohibited medicationsMedical conditions that would affect absorption, distribution, metabolism, or excretion of study treatment
* Unstable or inadequately treated medical
* An absolute neutrophil count (ANC) of ≤1.5 X 109 per liter
* Subject is pregnant or breastfeeding.
* Subject is taking other medication thought to directly affect gut function via the 5HT method of action (Tegaserod)
* Known hypersensitivity to duloxetine or any of the inactive ingredients in duloxetine
* Any patient taking Monoamine Oxidase Inhibitors
* Patient with uncontrolled narrow-angle glaucoma

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2008-02; Primary Completion 2012-01 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas A Drossman, MD, Principal Investigator — UNC Chapel Hill
Locations (1):
- UNC Center for Functional GI & Motility Disorders, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from UNC GI outpatient clinic. Other recruitment strategies like newspaper ads, UNC mass emails and flyers were used. Recruitment started around 12/2007.
Pre-assignment Details: This was 13 week long study which included 1 week of screning period followed by 4 weeks of treatment phase and 4 weeks of follow up period. During the screening visit following procedures were done- informed consent,medical history and demographics collection Vitals including abdominal girth,physical examination baseline labs and questionnaires
Groups:
- Quetiapine ( 50mg/Day -100mg/Day): There is only one group. All Subjects begin with a dose quetiapine of 50 mg for 2 weeks, increasing to 100 mg for the remainder of the study. 25 subjects were enrolled in this group.
Period: Overall Study
Arm/Group | Quetiapine ( 50mg/Day -100mg/Day)
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Subjects who received the investigational medication were analyzed. 4 subjects did not meet the study inclusion/exclusion criteria and were not analyzed.
Groups:
- Quetiapine ( 50mg/Day -100mg/Day): There is only one group. All Subjects begin with a dose quetiapine of 50mg for 2 weeks, increasing to 100 mg for the remainder of the study. (9 weeks total) 25 subjects were enrolled in this group.
Arm/Group | Quetiapine ( 50mg/Day -100mg/Day)
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.8 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Adequate Relief in Pain Score During Treatment
Description: Biweekly relief in pain Biweekly subjects were asked whether they had adequate relief of pain. It was binary questionnaire i.e.- " Did you have adequate relief of pain in last two weeks? 1) yes 2) no The measure is percentage of subjects who said yes who had adequate relief of pain.
Time Frame: 8 weeks
Population: There was no exact statistical test used to determine the sample size. It is based on the capacity of site to recruit subjects.
Measure: Number; unit: percentage of subjects
Groups:
- Quetiapine ( 50mg/Day -100mg/Day): There is only one group. All Subject begin with a dose quetiapine of 50mg for 2 weeks, increasing to 100 mg for the remainder of the study. (9 weeks total)30 subjects were enrolled in this group.
Arm/Group | Quetiapine ( 50mg/Day -100mg/Day)
Number analyzed (Participants) | 25
percentage of subjects | 52.6 (2.0)

ADVERSE EVENTS:
Time Frame: 3 years
Groups:
- Quetiapine ( 50mg/Day -100mg/Day): There is only one group. All Subject begin with a dose Quetiapine of 50 mg for 2 weeks, increasing to 100 mg for the remainder of the study. (9 weeks total)29 subjects were enrolled in this group.
Arm/Group | Quetiapine ( 50mg/Day -100mg/Day)
Serious Adverse Events (participants affected / at risk) | 1/25
Other Adverse Events (participants affected / at risk) | 23/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quetiapine ( 50mg/Day -100mg/Day) (N=25)
cerebrovascular accident (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quetiapine ( 50mg/Day -100mg/Day) (N=25)
Drowsiness (Nervous system disorders) | 23 (23)
tiredness (Musculoskeletal and connective tissue disorders) | 17 (17)
worsening abdominal pain or discomfort (Gastrointestinal disorders) | 4 (4)

LIMITATIONS AND CAVEATS:
1. Uncontrolled open label study and is vulnerable to biases favoring a treatment response.
2. Sample size is small.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No